CLINICAL TRIAL: NCT01809379
Title: Feasibility, Efficacy and Safety of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) With Cisplatin and Doxorubicin in Women With Recurrent Ovarian Cancer: an Open-label, Single-arm Phase II Clinical Trial
Brief Title: Intraperitoneal Aerosol High-pressure Chemotherapy for Women With Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Prof. Dr. med. Clemens Tempfer, MBA, Ruhr University of Bochum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIPAC-OV1
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Recurrent Ovarian Cancer
Keywords: ovarian cancer, recurrent, chemotherapy, intraperitoneal
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — Drug Therapy; Doxorubicin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intraperitoneal chemotherapy (Experimental): Intraperitoneal chemotherapy with cisplatin at a dose of 7.5 mg/m2 body surface in a 150 ml NaCl 0.9% and doxorubicin at a dose of 1.5 mg/m2 body surface in a 50 ml NaCl 0.9% solution with a flow of 30 ml/min and a max upstream pressure of 200 psi.
  Interventions: Drug: chemotherapy with doxorubicin and cisplatin

INTERVENTIONS:
Drug: chemotherapy with doxorubicin and cisplatin — intraperitoneal chemotherapy applied as an aerosol and under pressure
  Other Names: CISPLATIN Teva, Adrimedac

SUMMARY:
This trial aims to assess efficacy and safety of an intraperitoneal, aerosol, high-pressure chemotherapy in women with recurrent ovarian cancer

DETAILED DESCRIPTION:
This study aims to investigate the therapeutic efficacy of PIPAC using doxorubicin and cisplatin in women with recurrent ovarian cancer and disease progression with peritoneal carcinomatosis. The primary objective of this study is to determine the Clinical Benefit Rate (CBR) according to RECIST criteria after three cycles of PIPAC with cisplatin and doxorubicin.

ELIGIBILITY:
Inclusion Criteria:

* at least 2 lines of previous chemotherapy
* recurrent ovarian cancer
* patient is mobile
* informed consent

Exclusion Criteria:

* ileus
* necessity of parenteral nutrition

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate | 6 months
  The clinical benefit rate comprises complete remission, partial remission, and stable disease according to RECIST criteria.

SECONDARY OUTCOMES:
safety | 6 months
  left heart ejection fraction, neurological status, laparoscopy complications intraoperative, laparoscopy complications postoperative until hospital discharge, re-admission to hospital, death

OTHER OUTCOMES:
tumor apoptosis assessment, videolaparoscopy assessment of response, CA 125 assessment of response | 6 months
  various measures of response to therapy on the clinical, biochemical, and histological level

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Tempfer, MD, Principal Investigator — Runr University Bochum
Locations (1):
- Ruhr University Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Tempfer CB, Winnekendonk G, Solass W, Horvat R, Giger-Pabst U, Zieren J, Rezniczek GA, Reymond MA. Pressurized intraperitoneal aerosol chemotherapy in women with recurrent ovarian cancer: A phase 2 study. Gynecol Oncol. 2015 May;137(2):223-8. doi: 10.1016/j.ygyno.2015.02.009. Epub 2015 Feb 18. PMID 25701703